CLINICAL TRIAL: NCT03879473
Title: Influence of Peri-procedural Management of Direct Oral Anticoagulants on the Incidence of Pocket Hematoma in Patients Undergoing Cardiac Rhythm Device Implantation
Brief Title: Direct Oral Anticoagulant Management for Cardiac Device Implantation
Acronym: StimAOD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Necker Enfants Malades (Other)
Responsible Party: Principal Investigator, Anne-Céline MARTIN, Doctor, Institut Necker Enfants Malades
Other Study IDs: CV185-614
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Anticoagulant, Perioperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Each year, tens of thousands of cardiac rhythm devices including pacemaker (PM) or implantable cardioverter-defibrillator (ICD) are implanted in France. More than 25% of patients undergoing cardiac device implantation receive long-term anticoagulation therapy, that increases the incidence of pocket hematoma with potential serious consequences for patients. Although more and more patients receive direct oral anticoagulants (DOACs), limited data currently exist on the perioperative management of DOAC-treated patients undergoing cardiac device implantation and the optimal strategy remains unclear. Especially, the time of DOAC resumption after the procedure is controversial.

We hypothesize that the time of DOAC resumption is the main risk factor of bleeding event in DOAC-treated patients undergoing cardiac device implantation, that is to say that a delayed DOAC resumption > 48 hours following the procedure will reduce pocket hematoma incidence compared with an early resumption, ≤ 48 hours, without increasing thromboembolic events. We propose here an observational multicentre national study to find out the optimal strategy.

ELIGIBILITY:
Inclusion Criteria:

* receiving DOAC (apixaban, rivaroxaban, dabigatran) for stroke prevention in atrial fibrillation at least 5 days prior to enrolment
* undergoing a cardiac rhythm device implantation (implantation or replacement of PM (1 or 2 leads) and ICD (1or 2 leads) with or without cardiac-resynchronization therapy
* informed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * receiving DOAC (apixaban, rivaroxaban, dabigatran) for stroke prevention in atrial fibrillation at least 5 days prior to enrolment
  * undergoing a cardiac rhythm device implantation (implantation or replacement of PM (1 or 2 leads) and ICD (1or 2 leads) with or without cardiac-resynchronization therapy
  * informed
Sampling Method: Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
number of patients with clinically significant pocket hematoma | 30 +/- 5 days
  hematoma requiring reoperation, and/or resulting in prolongation of hospitalization, and/or requiring interruption of all anticoagulation.

SECONDARY OUTCOMES:
number of patients with thromboembolic event | 30 +/- 5 days
  transient ischemic attack, stroke, peripheral embolus, venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Céline Martin, MD, PhD, Principal Investigator — INSERM 1140
Locations (1):
- HEGP, Paris, France